CLINICAL TRIAL: NCT03575065
Title: An Open Label, Multi-Center Phase 2 Study to Evaluate Efficacy and Safety of BGB-290 in the Treatment of Metastatic HER2-Negative Breast Cancer Patients With BRCA Mutation in China
Brief Title: Efficacy and Safety of BGB-290 in the Treatment of Metastatic HER2-Negative Breast Cancer Patients With BRCA Mutation in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-201; CTR20171623 (Registry Identifier: National Medical Products Administration- NMPA)
Record Dates: First submitted 2018-06-19; First posted 2018-07-02 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: HER2-negative Breast Cancer
MeSH Terms: interventions — pamiparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Triple-negative breast cancer (TNBC) (Experimental): Locally advanced or metastatic TNBC
  Interventions: Drug: BGB-290
- Cohort 2: HR(+)/HER2(-) breast cancer (Experimental): Locally advanced or metastatic Hormone receptor-positive(HR+) human epidermal growth factor receptor2 Negative(HER2-) breast cancer
  Interventions: Drug: BGB-290

INTERVENTIONS:
Drug: BGB-290 — Administered orally
  Other Names: Pamiparib

SUMMARY:
This is a Phase 2, open-label, multi-center study of BGB-290 administered orally (PO) twice daily (BID) in adult Chinese patients with advanced HER2(-) breast cancer harboring germline BRCA mutation, which have progressed despite standard therapy, or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed deleterious or suspected deleterious germline BRCA1 or BRCA2 mutation
2. Locally advanced or metastatic breast cancer despite standard therapy and the following:

   1. Histologically or cytologically confirmed HER2(-) breast cancer (TNBC or estrogen receptor-positive and/or PR+)
   2. ≤ 2 prior lines of chemotherapy in advanced or metastatic setting
   3. Prior platinum therapy allowed as long as no disease progression while on treatment, or if given in neoadjuvant/adjuvant setting with ≥ 6 months from last platinum to relapse
   4. Prior therapy with an anthracycline and/or a taxane in neoadjuvant/adjuvant or metastatic setting
   5. Archival tumor tissues will be collected from all patients, if available
   6. For HR(+)/HER2(-) breast cancer only: patients must have received and progressed on at least one endocrine therapy either in adjuvant or metastatic setting, or have disease that the treating physician believes to be inappropriate for endocrine therapy
3. Measurable disease as defined per RECIST, version 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Adequate hematologic and organ function

Exclusion Criteria:

1. Unresolved acute effects of prior therapy of ≥ Grade 2
2. Prior treatment with a poly[ADP-ribose] polymerase (PARP) inhibitor
3. Chemotherapy, radiotherapy, biologic therapy, immunotherapy, investigational agent, anticancer Chinese medicine, or anticancer herbal remedies ≤ 14 days (or ≤ 5 half lives, if applicable, whichever is shorter) prior to Day 1 of Cycle 1
4. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 14 days prior to Day 1 of Cycle 1, or anticipation of need for major surgical procedure during the course of the study
5. Diagnosis of myelodysplastic syndrome (MDS)
6. Other diagnosis of malignancy
7. Untreated and/or active brain metastases.
8. Active infection requiring systemic treatment, active viral hepatitis, or active tuberculosis
9. Clinically significant cardiovascular disease
10. Pregnancy or nursing
11. Known history of intolerance to the excipients of the BGB-290 capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (20):
- China (20):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University Wuhan, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Xu B, Zhang QY, Yang H, Gu T, Zhang K, Liang J, Qiu JJ, Yang R, Zhang L, Mu S, Sun J, Huang V, Dong M. An Open-Label, Multicenter, Phase 2 Study to Evaluate the Antitumor Activity and Safety of Pamiparib in the Treatment of Metastatic HER2-Negative Breast Cancer Patients With BRCA Mutation in China. Chinese Society of Clinical Oncology. 2018.
- [Background] Xu B, Sun T, Shi Y, Cui J, Yin Y, Ouyang Q, Liu Q, Zhang Q, Chen Y, Wang S, Wang X, Tong Z, Zhong Y, Wang J, Yan M, Yan X, Wang C, Feng J, Wang X, Hu G, Cheng Y, Ge R, Zhu Z, Zhang W, Shao Z. Pamiparib in patients with locally advanced or metastatic HER2-negative breast cancer with germline BRCA mutations: a phase II study. Breast Cancer Res Treat. 2023 Feb;197(3):489-501. doi: 10.1007/s10549-022-06785-z. Epub 2022 Dec 2. PMID 36459284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 88 participants were recruited in China.
Groups:
- Triple-negative Breast Cancer (TNBC): Participants received 60 milligrams (mg) pamiparib twice daily (BID) orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
- Hormone Receptor-positive(HR+) Human Epidermal Growth Factor receptor2 Negative(HER2-) Breast Cancer: Participants received 60 mg pamiparib BID orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
Period: Overall Study
Arm/Group | Triple-negative Breast Cancer (TNBC) | Hormone Receptor-positive(HR+) Human Epidermal Growth Factor receptor2 Negative(HER2-) Breast Cancer
Started | 62 | 26
Completed | 0 | 0
Not Completed | 62 | 26
Not completed — Death | 31 | 12
Not completed — Sponsor's Decision | 28 | 13
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of pamiparib (BGB-290)
Groups:
- TNBC; HR(+)/HER2(-) Breast Cancer: Participants received 60 mg pamiparib BID orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
- Total: Total of all reporting groups
Arm/Group | TNBC | HR(+)/HER2(-) Breast Cancer | Total
Number analyzed (Participants) | 62 | 26 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (8.56) | 46.4 (10.75) | 45.8 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 26 | 88
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese | 62 | 26 | 88

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Independent Radiology Review (IRC)
Description: ORR is defined as the percentage of participants who achieved a best overall response of confirmed complete response (CR) or partial response (PR), assessed by IRC per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Time Frame: From the first dose of pamiparib to first documentation of disease progression while participant is alive (Approximately 2 years and 4 months)
Population: Efficacy Evaluable Analysis Set: includes all participants in the safety population who have measurable disease at baseline per RECIST v1.1 by IRC and have at least one evaluable post baseline tumor assessment by IRC unless discontinued treatment due to clinical progression or death prior to tumor assessment. Participants with available data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HR(+) /HER2(-) Breast Cancer: Participants received 60 mg pamiparib BID orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 55 | 21
Percentage of participants | 38.2 [25.4 to 52.3] | 61.9 [38.4 to 81.9]
Statistical Analysis 1: Comparison: TNBC; Test type: Superiority; p = 0.0210, Exact Binomial Test — p-value was based on an exact binomial test with historic control ORR=0.25

2. Secondary Outcome: ORR as Assessed by Investigator
Description: ORR is defined as the percentage of participants who achieved a best overall response of confirmed complete response (CR) or partial response (PR), assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Time Frame: From the first dose of pamiparib to first documentation of disease progression while participant is alive (Approximately 2 years and 10 months)
Population: Efficacy Evaluable Analysis Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 55 | 21
Percentage of participants | 36.4 [23.8 to 50.4] | 57.1 [34.0 to 78.2]

3. Secondary Outcome: Progression-free Survival (PFS) as Assessed by IRC and Investigator
Description: PFS is defined as the time from first dose of pamiparib to the first documented disease progression or death due to any cause, assessed by IRC or the investigator
Time Frame: From the first dose of pamiparib to first documentation of disease progression or death (Approximately 2 years and 10 months)
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 62 | 26
Months
  IRC | 5.49 [3.65 to 7.33] | 9.20 [7.39 to 11.93]
  Investigator | 3.78 [3.68 to 6.41] | 9.69 [5.55 to 12.85]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by IRC
Description: DOR is defined as the time from first determination of a confirmed best overall response until the first documentation of progression or death, whichever comes first, assessed by IRC
Time Frame: From first documentation of confirmed CR or PR to first documentation of disease progression or death (Approximately 2 years and 10 months)
Population: Efficacy Evaluable Analysis Set; Only the participants with confirmed objective responses by IRC were included in DOR analysis;
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 21 | 13
Months | 6.97 [3.94 to NA] — NA = NE Not estimable due to insufficient number of events | 7.49 [5.55 to 14.75]

5. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator
Description: DOR is defined as the time from first determination of a confirmed best overall response until the first documentation of progression or death, whichever comes first, assessed by the investigator
Time Frame: as for outcome 4
Population: Efficacy Evaluable Analysis Set; Only the participants with confirmed objective responses by Investigator were included in DOR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 20 | 12
Months | 6.28 [4.63 to 11.76] | 11.57 [5.95 to 13.90]

6. Secondary Outcome: Confirmed Best Overall Response (BOR) as Assessed by IRC and Investigator
Description: BOR is defined as the percentage of participants with best overall response recorded from the start of the treatment until disease progression or recurrence, assessed by IRC or the investigator. BOR included complete response [CR], partial response [PR], stable disease [SD], disease progression and not evaluable [NE].
Time Frame: Approximately 2 years and 10 months
Population: Efficacy Evaluable Analysis Set; Participants with available data were included in the analysis
Measure: Number; unit: Percentage of participants
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 55 | 21
Percentage of participants
  IRC - CR | 5.5 | 4.8
  IRC - PR | 32.7 | 57.1
  IRC - SD | 34.5 | 28.6
  IRC - PD | 27.3 | 9.5
  IRC - NE | 0 | 0
  Investigator - CR | 3.6 | 0
  Investigator - PR | 32.7 | 57.1
  Investigator - SD | 36.4 | 23.8
  Investigator - PD | 27.3 | 19.0
  Investigator - NE | 0 | 0

7. Secondary Outcome: Disease Control Rate (DCR) as Assessed by IRC and Investigator
Description: DCR is defined as the percentage of participants who achieved a confirmed BOR of CR, PR, or stable disease (SD), assessed by IRC or the investigator
Time Frame: as for outcome 2
Population: Efficacy Evaluable Set; Participants with available data were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 55 | 21
Percentage of participants
  IRC | 72.7 [59.0 to 83.9] | 90.5 [69.6 to 98.8]
  Investigator | 72.7 [59.0 to 83.9] | 81.0 [58.1 to 94.6]

8. Secondary Outcome: Clinical Benefit Rate (CBR) as Assessed by IRC and Investigator
Description: CBR is defined as percentage of participants with confirmed CR or confirmed PR or a durable SD (SD lasting ≥ 24 weeks), assessed by IRC or the investigator
Time Frame: as for outcome 2
Population: Efficacy Evaluable Set; Participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 55 | 21
Percentage of participants
  IRC | 43.6 [30.3 to 57.7] | 71.4 [47.8 to 88.7]
  Investigator | 41.8 [28.7 to 55.9] | 66.7 [43.0 to 85.4]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the first dose of pamiparib to the date of death due to any cause
Time Frame: From the first dose of pamiparib until death (approximately 2 years and 10 months)
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TNBC | HR(+) /HER2(-) Breast Cancer
Number analyzed (Participants) | 62 | 26
Months | 17.08 [15.57 to NA] — NA = NE Not estimable due to insufficient number of events | 27.89 [18.10 to NA] — NA = NE Not estimable due to insufficient number of events

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: A TEAE is defined as an adverse event (AE) that had an onset date on or after the first dose of study drug up to 30 days following study drug discontinuation. SAE is defined as any AE that leads to death or is life-threatening.
Time Frame: Up to approximately 2 years and 10 months
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- HR(+) / HER2(-) Breast Cancer: Participants received 60 mg pamiparib BID orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
Arm/Group | TNBC | HR(+) / HER2(-) Breast Cancer
Number analyzed (Participants) | 62 | 26
participants
  With At Least 1 TEAE | 61 | 26
  Grade 3 or higher | 37 | 18
  SAEs | 12 | 7

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years and 10 months
Groups:
- HR(+)/HER2(-): Participants received 60 mg pamiparib BID orally in 28-day cycles until disease progression, unacceptable toxicity, death, withdrawal of consent or study termination by sponsor
Arm/Group | TNBC | HR(+)/HER2(-)
All-Cause Mortality (participants affected / at risk) | 31/62 | 12/26
Serious Adverse Events (participants affected / at risk) | 12/62 | 7/26
Other Adverse Events (participants affected / at risk) | 61/62 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNBC (N=62) | HR(+)/HER2(-) (N=26)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNBC (N=62) | HR(+)/HER2(-) (N=26)
Anaemia (Blood and lymphatic system disorders) | 51 (79) | 26 (40)
Leukopenia (Blood and lymphatic system disorders) | 8 (20) | 6 (15)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (7) | 3 (7)
Neutropenia (Blood and lymphatic system disorders) | 5 (15) | 5 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (41) | 15 (35)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (32) | 14 (30)
Asthenia (General disorders) | 9 (10) | 4 (4)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (5)
Influenza like illness (General disorders) | 2 (2) | 2 (2)
Malaise (General disorders) | 11 (11) | 4 (4)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 6 (10)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 13 (17) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 10 (13) | 7 (7)
Bilirubin conjugated increased (Investigations) | 3 (4) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 6 (8)
Blood bilirubin increased (Investigations) | 8 (10) | 7 (8)
Blood bilirubin unconjugated increased (Investigations) | 2 (3) | 4 (5)
Blood creatinine increased (Investigations) | 1 (1) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 4 (5) | 2 (2)
Lipoprotein (a) increased (Investigations) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 2 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (8) | 1 (2)
Neutrophil count decreased (Investigations) | 34 (111) | 18 (28)
Platelet count decreased (Investigations) | 19 (28) | 11 (11)
Weight decreased (Investigations) | 11 (14) | 1 (1)
Weight increased (Investigations) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 35 (132) | 21 (35)
Decreased appetite (Metabolism and nutrition disorders) | 25 (28) | 8 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 3 (6)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (7) | 5 (7)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03575065/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03575065/SAP_001.pdf